CLINICAL TRIAL: NCT03303222
Title: Pilot Study to Develop a Breath Analyser to Detect Chronic Kidney Disease
Brief Title: Study to Develop a Breath Analyser to Detect Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 228416
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients on dialysis: patients with kidney disease treated by dialysis
  Interventions: Diagnostic Test: breath
- patients with chronic kidney disease: patients with chronic kidney disease not treated by dialysis
  Interventions: Diagnostic Test: breath

INTERVENTIONS:
Diagnostic Test: breath — measurement of volatile compounds, such as TMAO in exhaled breath and blood
  Other Names: blood sample

SUMMARY:
Measure trimethylamine oxide in the breath.

DETAILED DESCRIPTION:
Organic compounds such as trimethylamine oxide (TMAO) accumulate in the blood of patients with kidney disease, and volatile compounds such as TMAO can be detected in the breath.

The investigators wish to develop a breath analyser to measure volatile compounds, such as TMAO in the breath in patients with kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with kidney disease under the care of Royal Free Hospital

Exclusion Criteria:

* patients unable to provide informed consent
* patients unable to exhale into breath analyser

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with kidney disease under the care of Royal Free Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-10 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
measurement of breath TMAO | 3 years
  measurement of breath TMAO by breath analyser

CONTACTS AND LOCATIONS:
Overall Officials: andrew davenport, md, Principal Investigator — UCL, London

IPD SHARING:
Plan to Share IPD: No
Data will be filed in UCL library as PhD submission